CLINICAL TRIAL: NCT06057597
Title: Randomized Controlled Non-inferiority Trial Evaluating the Safety and Efficacy of the Omega Gastric Bypass With 150 cm Biliopancreatic Loop Length Compared to the Roux-en-Y Gastric Bypass
Brief Title: Omega Gastric Bypass (150cm) Compared to the Roux-en-Y Gastric Bypass (YOMEGA-2 Multicentric Trial)
Acronym: YOMEGA-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP211050
Record Dates: First submitted 2023-04-03; First posted 2023-09-28 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Morbid
Keywords: Bariatric surgery; RYGB; MGB/OAGB
MeSH Terms: conditions — Obesity | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): This corresponds to patients with type 2 obesity (BMI 35-40) with comorbidities (high blood pressure, type 2 diabetes mellitus, obstructive sleep apnea, dyslipidemia, arthrosis) and type 3 obesity (BMI ≥ 40 kg/m²) and candidates for bariatric surgery.
  Laparoscopic OAGB will be performed with long and narrow gastric pouch (30cc) and 150 cm biliopancreatic limb
  Interventions: Procedure: Laparoscopic OAGB
- Control Groupe (Active Comparator): This corresponds to patients with type 2 obesity (BMI 35-40) with comorbidities (high blood pressure, type 2 diabetes mellitus, obstructive sleep apnea, dyslipidemia, arthrosis) and type 3 obesity (BMI ≥ 40 kg/m²) and candidates for bariatric surgery.
  Standard laparoscopic RYGB will be performed with a gastric pouch (30cc) and 150 cm antecolic Roux limb and a 50 cm biliopancreatic limb.
  Interventions: Procedure: Laparoscopic RYGB

INTERVENTIONS:
Procedure: Laparoscopic OAGB — It is a gastric bypass surgery with a unique gastro-jejunal anastomosis, a long (11-14cm) and narrow (3-4cm) gastric pouch will be created by applying one horizontal 45-mm stapler at the angle of lesser curvature, just above the left branch of the crow's foot, and then four to five vertical 60-mm staple cartridges will be placed upwards to the angle of His, and calibrated along a 32-Fr bougie. Sectioning of the greater omentum into a bivalve will be performed. The jejunum will be measured using pre-measured strip and amounted antecolically at 150 cm from the ligament of Treitz. An end-to-side anastomosis will be performed with the gastric pouch, using a 45-mm linear stapler and an anterior running suture to close gastro-enterotomy.
  Other Names: One Anastomosis Gastric Bypass / Mini Gastric Bypass
  Arms: Experimental group
Procedure: Laparoscopic RYGB — A small gastric pouch (30cc) will be created using a linear stapler. The alimentary limb will be moved up into an antecolic position after an epiploic transection so as to perform the gastro-jujunal anastomosis. The gastro-jejunostomy will be performed manually or using a linear or circular stapler. An alimentary limb of 150 cm and a biliary limb of 50cm will be measured (using premeasured strip) in order to perform the latero-lateral jejuno-jejunal anastomosis using a linear stapler. All mesenteric defects (Petersen's space and mesenteric defect) will be closed with a non-absorbable running suture
  Other Names: Roux-en-Y Gastric Bypass
  Arms: Control Groupe

SUMMARY:
Obesity with its consequences such as type 2 diabetes, high blood pressure, dyslipidemia, fatty liver disease, sleep apnea and cancers, remains a major healthcare problem worldwide. Bariatric surgery, combined with nutritional education and close monitoring, has been shown to be the most effective treatment for patients with morbid obesity resulting in significant and lasting weight loss and improvements in co-morbidities . With nearly 50000 procedures per year France ranks third in the world in terms of care for patients suffering from morbid (BMI ≥ 40 kg/m²) and severe (BMI 35-40 kg/m²) obesity.

In parallel with the significant increase in the number of patients operated on for obesity in the world, over the past two decades, significant development has been observed in the field of bariatric surgery with a decrease or even disappearance of some procedures and the appearance of others.

Performed for more than 40 years, the Roux-en-Y Gastric Bypass (RYGB) is a restrictive and malabsorptive procedure and currently is considered as gold standard procedure for the treatment of morbid obesity and its comorbidities. However, despite the good effectiveness (with an average Excess Weight Loss % (EWL%) of approximatively 70% at 2 years), RYGB is technically demanding procedure with learning curve requiring more than 100 cases and an overall complication rate ranging from 10% to 20% Introduced in 2001, one anastomosis gastric bypass (OAGB) is a modified gastric bypass that consists of a single gastrojejunal anastomosis between a long gastric pouch and a jejunal (biliopancreatic) omega loop. In Sept. 2019, taking into account the results from YOMEGA trial, the French High Authority for Health (Haute Autorité de Santé (HAS)) recommended to ban OAGB with 200 cm or longer BPL and urged to assess the efficacy and safety of OAGB with 150 cm BPL in a randomized controlled trial. Indeed, YOMEGA-2 trial is logical continuity of the YOMEGA trial.

The aim of this study is to assess weight loss efficiency and the nutritional safety of the OAGB-150 in comparison to a standard (RYGB).

The hypothesis of this study is that the OAGB with a 150 cm BPL could have the same efficacy on weight loss and nutritional complication rate in comparison to the RYGB at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged from 18 to 65 years old
* Type III obesity (BMI ≥ 40 kg/m²), or Type II obesity BMI 35-40 kg/m2 associated with at least one co-morbidity which will be improved by surgery (high blood pressure, type 2 diabetes mellitus, obstructive sleep apnea, dyslipidemia, arthrosis)
* Patient who had benefited from an Upper GI Endoscopy with biopsies to look for Helicobacter pylori within 12 months before surgery
* Patient who has benefited from a multidisciplinary evaluation at least 6 months, with a favorable opinion for a gastric bypass
* Patient who understood and accepted the need for a long-term follow-up
* Patient who agreed to be included in the study and who signed the informed consent form
* Patient affiliated to a social security scheme
* For child-bearing aged women, efficient contraception

Exclusion Criteria:

* History of previous bariatric surgery
* History of chronic inflammatory bowel disease
* Presence of chronic diarrhea
* Presence of a severe and evolutive life threatening pathology
* Presence of dysplastic modifications of the gastric mucosa, chronic atrophic gastritis or history of gastric cancer
* Presence of an unhealed gastro-duodenal ulcer
* Presence of Helicobacter pylori resistant to medical treatment
* Presence of esophagitis
* Pregnancy or desire to be pregnant during the study
* Mentally unbalanced patients, under supervision or guardianship
* Patients who don't understand French and not able to give consent
* Patient included and followed in another interventional trial
* Unable to consent, under tutelage or curatorship, or judiciary safeguard

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
To demonstrate that OAGB with 150 cm biliopancreatic limb is not inferior to RYGB on weight loss (efficacy). | 2 years after the surgery
  For each patient co-primary endpoints will be assessed at 2 years after surgery composed by:
  Efficacy: Weight loss according to Excess Weight Loss % (EWL%) calculated using the following formula: ((weight 2 years after surgery - initial weight) / (initial weight - ideal weight)) x 100. Ideal weight defined as the weight corresponding to a BMI = 25 kg/m².
  The assessment of the primary co-endpoint will be standardized between the sites.
To demonstrate that OAGB with 150 cm biliopancreatic limb is not inferior to RYGB on nutritional complication rate (safety) | 2 years after the surgery
  For each patient co-primary endpoints will be assessed at 2 years after surgery composed by:
  Safety: Nutritional complications defined by at least one vitamin deficiency (vit. B1 < 66nmol/l or B12 < 145pmol/l), malnutrition (albumin < 30g/l), anemia (hemoglobin < 10g/dl) or a combination of these.
  The assessment of the primary co-endpoint will be standardized between the sites.

SECONDARY OUTCOMES:
Measurement of albumin | Before and 1, 3, 6, 12, 18 and 24 months after surgery
  Measurement of albumin will explore the nutritional status of patients. Results will be expressed in g/l
Measurement of pre-albumin | Before and 1, 3, 6, 12, 18 and 24 months after surgery
  Measurement of pre-albumin will explore the nutritional status of patients. Results will be expressed in g/l
Measurement of hemoglobin | Before and 1, 3, 6, 12, 18 and 24 months after surgery
  Measurement of hemoglobin will explore the nutritional status of patients. Results will be expressed in g/l
Measurement of calcium | Before and 1, 3, 6, 12, 18 and 24 months after surgery
  Measurement of calcium will explore the nutritional status of patients. Results will be expressed in mmol/l
Measurement of ferritin | Before and 1, 3, 6, 12, 18 and 24 months after surgery
  Measurement of ferritin will explore the nutritional status of patients. Results will be expressed in μg/l
Measurement of iron | Before surgery and 1, 3, 6, 12, 18 and 24 months after surgery
  Measurement of iron will explore the nutritional status of patients. Results will be expressed in mmol/l
Measurement of % of transferrin saturation | Before surgery and 1, 3, 6, 12, 18 and 24 months after surgery
  Measurement of % of transferrin saturation will explore the nutritional status of patients. Results will be expressed in %
Measurement of zinc | Before surgery and 6, 12 months and 24 months after surgery
  Measurement of zinc will explore the nutritional status of patients. Results will be expressed in mmol/L
Measurement of vitamin A | Before surgery and 6, 12 and 24 months after surgery
  Measurement of vitamin A will explore the nutritional status of patients. Results will be expressed in mmol/l
Measurement of vitamin B1 | Before surgery and 6, 12 and 24 months after surgery
  Measurement of vitamin B1 will explore the nutritional status of patients. Results will be expressed in nmol/l
Measurement of vitamin B9 | Before surgery and 6, 12 and 24 months after surgery
  Measurement of vitamin B9 will explore the nutritional status of patients. Results will be expressed in nmol/l
Measurement of vitamin B12 | Before surgery and 6, 12 and 24 months after surgery
  Measurement of vitamin B12 will explore the nutritional status of patients. Results will be expressed in pmol/l
Measurement of vitamin E | Before surgery and 6, 12 and 24 months after surgery
  Measurement of vitamin E will explore the nutritional status of patients. Results will be expressed in mmol/l
Measurement of vitamin D | Before surgery and 6, 12 and 24 months after surgery
  Measurement of vitamin D will explore the nutritional status of patients. Results will be expressed in nmol/l
Measurement of prothrombin rate | Before surgery and 6, 12 and 24 months after surgery
  Measurement of prothrombin rate will explore the nutritional status of patients. Results will be expressed in %
Measurement of the 24-hour steatorrhea rate | 6 month after surgery
  Measurement of the average number of stool will explore the nutritional status of patients. Results will be expressed in number of stool/day
Measurement of HbA1c | Before surgery and 1, 3, 6, 12, 18 and 24 months after surgery
  Measurement of HbA1c will explore the Metabolic efficiency of surgery. Results will be expressed in %
Measurement of fasting glycemia | Before surgery and 1, 3, 6, 12, 18 and 24 months after surgery
  Measurement of fasting glycemia will explore the Metabolic efficiency of surgery. Results will be expressed in mmol/l
Measurement of HDL | Before surgery and 1, 3, 6, 12, 18 and 24 months after surgery
  Measurement of HDL will explore the Metabolic efficiency of surgery. Results will be expressed in mmol/l
Measurement of LDL | Before surgery and 1, 3, 6, 12, 18 and 24 months after surgery
  Measurement of LDL will explore the Metabolic efficiency of surgery. Results will be expressed in mmol/l
Measurement of cholesterol | Before surgery and 1, 3, 6, 12, 18 and 24 months after surgery
  Measurement of cholesterol will explore the Metabolic efficiency of surgery. Results will be expressed in mmol/l
Measurement of triglycerides | Before surgery and 1, 3, 6, 12, 18 and 24 months after surgery
  Measurement of triglycerides will explore the Metabolic of surgery. Results will be expressed in mmol/l
Evaluation of antidiabetic drugs | Before surgery and 6, 12 and 24 months after surgery
  Assessment of number of antidiabetic medications will explore the Metabolic efficiency of surgery. This outcome will be expressed in terms of increase, decrease, discontinuation or restart of treatment.
Evaluation of antilipidemic drugs | Before surgery and 6, 12 and 24 months after surgery
  Assessment of the number of antilipidemic medications will explore the Metabolic efficiency of surgery. This outcome will be expressed in terms of increase, decrease, discontinuation or restart of treatment
Evaluation of antihypertensive drugs | Before surgery and 6, 12 and 24 months after surgery
  Assessment of the number of antihypertensive medications will explore the Metabolic efficiency of surgery. This outcome will be expressed in terms of increase, decrease, discontinuation or restart of treatment.
Evaluation of the use of Continuous Positive Airway Pressure for Obstructive Sleep Apnea | Before surgery and 6, 12 and 24 months after surgery
  Evolution of the use of Continuous Positive Airway Pressure for Obstructive Sleep Apnea will explore the Metabolic efficiency of surgery. This outcome will be expressed in terms of the use or discontinuation of the use of Continuous Positive Airway Pressure machine
Hospitalization length | The last day of hospitalization
  The Length of stay (in days) is based on the number of days of hospitalization from surgery (day of surgery = D0) until the end of hospitalization.
Number of patients readmitted | 30 days after surgery
  Number of patients readmitted within 30 days after surgery.
Occurrence of kidney stone | Within 2 years after surgery
  For each visit after the surgery, the presence or not of kidney stones will be documented and if applicable the treatment will be noted
Overall complications rate | Within 24 months after surgery
  Rate of medical and surgical (> or = grade III) complications within 24 months after surgery using the Dindo-Clavien classification, described as :
  Grade I = Any deviation from the normal postoperative course. Grade II = Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Grade III = Requiring surgical, endoscopic or radiological intervention, not under (Grade IIIa) or under general anesthesia (Grade IIIb) Grade IV = Life-threatening complication with single organ (Grade IVa) or Multiorgan dysfunction (Grade IVb) Grade V = Death of a patient.
Type of early complications | Within 30 days after surgery
  Type (medical or surgical) of early complications (within 30 days) for each procedure.
Severity of early complications | Within 30 days after surgery
  Severity of early complications (within 30 days) for each procedure according to the Dindo-Clavien classification
Type of late complications | Within 2 years after surgery
  Type (medical or surgical) of late complications (after 30 days) for each procedure.
Severity of late complications | Within 2 years after surgery
  Severity of late complications (after 30 days) for each procedure according to the Dindo-Clavien classification
Gastroesophageal reflux assessment | Before surgery and 1, 3, 6, 12, 18 and 24 months after surgery
  Evolution of gastroesophageal reflux will be assessed at each study visit, before and after surgery. This outcome will be expressed in terms of improvement, aggravation or onset.
Absolute weight loss assessment | 1, 3, 6, 12, 18 and 24 months after surgery
  Weight loss at 1, 3, 6, 12, 18 and 24 months after surgery, according to absolute weight loss (aWL) in kg.
Excess Weight Loss percentage assessment | 1, 3, 6, 12, 18 and 24 months after surgery
  Weight loss at 1, 3, 6, 12, 18 and 24 months after surgery, according to Excess Weight Loss percentage (EWL%), calculated using the following formula:
  ((weight at visit X - initial weight) / (initial weight - ideal weight)) X 100
Excess BMI Loss percentage assessment | 1, 3, 6, 12, 18 and 24 months after surgery
  Weight loss at 1, 3, 6, 12, 18 and 24 months after surgery, according Excess BMI Loss percentage (EBL%), according to the formula :
  ((BMI at visit X - initial BMI) / (initial BMI - ideal BMI)) X 100 with Ideal BMI = 25 kg/m²
Quality of life assessed with GIQLI questionnaire | Before surgery and at 6, 12 and 24 months after surgery
  This questionnaire consists of 36 items exploring 5 dimensions or subscales: symptoms, physical condition, emotions, social integration and the effect of any medical treatment. For each item, 5 responses will be proposed to the patients and for each answer, a score ranging from 0 to 4 (highest score = 144) will be assigned. A high score defines a more favorable health state
Quality of life assessed with SF36 questionnaire | Before surgery and at 6, 12 and 24 months after surgery
  This questionnaire taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/tiredness, and general health perceptions. It also includes a single item that provides an indication of a perceived change in health
Quality of life assessed with Sigstad questionnaire | Before surgery and at 1, 3, 6, 12, 18 and 24 months after surgery
  The Sigstad questionnaire allows the identification and diagnosis of postoperative dumping syndrome and early hypoglycaemia: a score >7 suggests a dumping syndrome
Body composition | Before and 24 months after surgery.
  Body composition level on a subsample of the total population:
  By impedancemetry :
  * Muscle mass index in kg/m2
  * Non-fat mass index in kg/m2
  * Fat mass index in kg/m2
Sarcopenia level | Before and 24 months after surgery.
  Sarcopenia level on a subsample of the total population will be assessed by Handgrip Strength

CONTACTS AND LOCATIONS:
Overall Officials: Tigran POGHOSYAN, MD-PhD, Principal Investigator — Bichat (APHP)
Locations (1):
- Hôpital Bichat Claude-Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: No